CLINICAL TRIAL: NCT06794957
Title: A Single-Arm, Open, Phase Ib Study Evaluating the Safety, Preliminary Efficacy of AL8326 in the Treatment of Non-Small Cell Lung Cancer
Brief Title: A Study of AL8326 in Non-Small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Advenchen Laboratories, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AL8326-CN-008
Record Dates: First submitted 2024-01-30; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-02

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- AL8326 (Experimental): Subject will received AL8326 once daily for 28-days cycle until intolerable toxicity or disease progression or death or voluntary withdrawal the end of this study. Subjects will be evaluated for anti-tumor efficacy and corresponding safety examinations every 2 cycles, and tumor disease status will be according to Response Evaluation Criteria in Solid Tumours（RECIST 1.1）.
  Interventions: Drug: AL8326 tablets

INTERVENTIONS:
Drug: AL8326 tablets — 10mg/tablet;Oral administration, once daily.
  Other Names: AL8326

SUMMARY:
This trial is a multicenter, single arm, open, phase IB clinical trial, designed to evaluate the preliminary efficacy and safety of AL8326 in patients with non-small cell lung cancer (NSCLC) who relapsed or progressed after multi line treatment and failed standard treatment.

DETAILED DESCRIPTION:
The subjects received the test drug al8326 tablets in the order of enrollment (oral administration, once a day, one cycle every 28 days) until intolerable toxicity or disease progression or death or voluntary withdrawal or the end of this study. The subjects will conduct anti-tumor efficacy evaluation and corresponding safety inspection every 2 cycles, and determine the tumor disease status according to the solid tumor efficacy evaluation criteria (RECIST 1.1).

Subjects requiring pharmacokinetic analysis will be randomly treated with trial drug AL8326 tablets 60mg QD or 40mg QD (oral administration, once a day, one cycle every 28 days) in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be able to understand and be willing to sign a written informed consent form before beginning any study-related procedures;
2. Age ≥18 years, both male and female;
3. Patients with advanced non-small cell lung cancer who failed standard treatment confirmed by pathology (disease progression after treatment or intolerable toxic and side effects of treatment) or did not have standard treatment (group A: Patients with non-small cell lung cancer without brain metastasis confirmed by imaging at baseline; group B: Patients with non-small cell lung cancer with brain metastasis confirmed by imaging at baseline)；
4. Have received at least two or more systemic treatment regimens;
5. Have at least one measurable tumor lesion according to the criteria for evaluating the efficacy of solid tumors (RECIST 1.1);
6. Have received prior chemotherapy with a cytotoxic agent, with an interval of at least 4 weeks between the end of chemotherapy and the time of enrollment, and have recovered to grade ≤1 (except alopecia areata) from a toxic reaction to prior chemotherapy
7. Life expectancy ≥ 12 weeks.
8. Eastern Cooperative Oncology Group（ECOG） score of 0 -1.
9. Subjects have adequate organ and bone marrow function and meet the following laboratory test criteria:

   1. Bone marrow function: absolute neutrophil count (ANC) ≥ 1.5 x 10^9 /L (1500/mm^3), platelets ≥ 80 x 10^9/L;cifang
   2. Hemoglobin ≥ 9.0 g/dl;
   3. Liver function: serum total bilirubin ≤ 1.5 times the upper limit of normal (ULN), except for patients with Gilbert's syndrome (persistent or recurrent hyperbilirubinemia manifesting as elevated unconjugated bilirubin in the absence of evidence of hemolysis or hepatic pathology); and for those without liver transfer, alanine aminotransferase ( ALT ）and aspartate aminotransferase (AST) ≤ 2.5 × ULN for those without liver metastases, and ALT and AST ≤ 5 × ULN for those with liver metastases;
   4. Renal function: serum creatinine ≤1.5×ULN and standardized endogenous creatinine clearance ≥60 ml/min estimated by the Cockcroft-Gault formula, Ccr(ml/min)=[(140-age)×body weight(kg)]/[72×Scr(mg/dl)], and for females, it is calculated as follows×0.85;
   5. Coagulation function: International Normalized Ratio (INR) ≤1.5;
   6. Screening period left ventricular ejection fraction (LVEF) > 50%.
10. Systolic blood pressure (SBP) < 140 mmHg and diastolic blood pressure (DBP) < 90 mmHg (no therapeutic drugs or single drug controllable).

11.1) Female: For female subjects of childbearing potential, they must have a negative serum pregnancy test within 7 days prior to enrollment and be using a medically licensed method of contraception during and for 3 months after completion of treatment; they must have a negative serum or urine pregnancy test during the Screening Period; they must not be breastfeeding; and they are considered to be of childbearing potential if they are menopausal but have not yet attained a postmenopausal status (menopausal for a period of time greater than or equal to 12 consecutive months for no reason other than no reason other than menopause) and has not undergone sterilization (removal of ovaries and/or uterus), such females are considered to be of childbearing potential. Their sexual partner is using a medically licensed method of contraception during and for 3 months after the end of the subject's treatment; 2) Males: surgical sterilization or medically licensed contraception during and for 3 months after the end of treatment; and their sexual partner is using a medically licensed method of contraception during and for 3 months after the end of the subject's treatment.

12.Ability and willingness to comply with study protocol requirements during the study and follow-up procedures.

Exclusion Criteria:

1. The patient used AL8326 tablets.
2. Allergic to AL8326 or its analogues, or to any component in the prescription of AL8326;
3. The last dose of systemic cytotoxic or investigational therapy was administered within 28 days prior to initiation of study treatment. Or the last dose of a non-cytotoxic, non-investigational treatment (i.e., radiation therapy, hormone therapy, targeted therapy, immunotherapy, etc.) was administered within 14 days prior to initiation of study treatment;
4. Major surgery (defined as requiring general anesthesia within 28 days prior to initiation of study treatment or general anesthesia for minor surgical procedures within 7 days prior to initiation of study treatment).
5. Pregnant or lactating female patients.
6. History of a prior or concurrent second primary malignancy that, in the opinion of the investigator or sponsor, may interfere with the assessment of the safety or efficacy of the investigational therapeutic agents.
7. Patients with active or untreated central nervous system（CNS） metastases; subjects with stabilized brain metastases will need to meet the following criteria for enrollment: a) no imaging-proven progression ≥4 weeks after completion of treatment; b) completion of treatment within ≥28 days prior to the first dose of the test drug; and c) no need to be treated with systemic corticosteroids (>10 mg/day of prednisone or equivalent dose) ≤28 days prior to the first dose of the test drug.
8. Peptic ulcer disease, inflammatory bowel disease, ulcerative colitis, or other gastrointestinal disease with risk of perforation; history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days prior to starting study treatment.
9. The patients have had an arterial/venous thrombotic event such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis and pulmonary embolism within 6 months prior to screening;
10. Presence of uncontrolled infection (within 2 weeks prior to administration of test drug).
11. New York Heart Association (NYHA) class III or IV congestive heart failure as achieved by cardiac function.
12. Had the following history of heart disease within 6 months before starting study treatment:

    1. Cardiac angioplasty or stenting, or
    2. Myocardial infarction, or
    3. Unstable angina, or
    4. Cerebrovascular accident
13. Imaging showed that the tumor had invaded around important blood vessels, or the investigator judged that the tumor was very likely to invade important blood vessels during the follow-up study and cause fatal massive hemorrhage;

15.With ascites or uncontrollable pleural effusion (CTCAE 5.0 ≥ grade 2). 16.Evidence of hemorrhagic idiosyncrasies or coagulation disorders or clinically significant bleeding (such as gross hematuria, gastrointestinal bleeding, and hemoptysis) detected within 6 months prior to initiation of study treatment.

17.Patients treated with anticoagulants or vitamin K antagonists (such as warfarin, heparin, or their analogues); Under the premise that the international standardized ratio of prothrombin time (INR) is ≤ 1.5, it is allowed to use low-dose anticoagulants for preventive purposes, such as warfarin (no more than 1mg per day, oral), low-dose heparin (no more than 12000 U per day), or low-dose aspirin (no more than 100mg per day); 18.There are arrhythmias that need clinical intervention (such as long QT syndrome, QTc corrected by fridericia formula is not measurable or > 450 ms in men and > 470 MS in women); 19.Within 28 days before starting the study treatment, urine protein was ≥ + +, and 24-hour urine protein quantitation was > 1.0g; 20.Hepatitis B surface antigen is positive and hepatitis B virus load (HBV-DNA) is higher than the lower limit of local laboratory detection, anti hepatitis C antibody is positive and hepatitis C virus load (HCV-RNA) is higher than the lower limit of local laboratory detection, Treponema pallidum antibody is positive, and human immunodeficiency virus anti physical examination result is positive.

21.History of organ transplantation. 22.Clinical symptoms affecting the intake or absorption of AL8326 (such as inability to swallow, chronic diarrhea, intestinal obstruction, malabsorptive disease, total gastrectomy or small bowel resection); 23.Prohibited combination drug therapy within 14 days prior to initiation of study treatment.

24.Red blood cell or platelet transfusion within 14 days prior to initiation of study treatment.

25.Any serious and/or unstable pre-existing medical, psychiatric, or other condition that may jeopardize the subject's safety, obtaining informed consent, or compliance with study procedures or study objectives.

26.Any other reason that, in the judgment of the investigator, makes participation in this study inappropriate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2022-05-19 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Objective remission rate (ORR) | Every 2 cycles,up to 24 months (each cycle is 28 days)
  The proportion of subjects achieving complete remission (CR) and partial remission (PR) with optimal efficacy according to RECIST 1.1.

SECONDARY OUTCOMES:
Duration of remission (DOR) | Every 2 cycles,up to 24 months (each cycle is 28 days)
  The time between the start of the first assessment of the tumor as CR or PR and The first assessment of disease progression (PD) or death from any cause.
Disease Control Rate (DCR) | Every 2 cycles,up to 24 months (each cycle is 28 days)
  The proportion of subjects achieving complete remission (CR), partial remission (PR) and stable disease (SD).
Duration of Disease Control (DDC) | Every 2 cycles,up to 24 months (each cycle is 28 days)
  The time from the first assessment of the tumor as CR, PR, or SD to the first assessment of disease progression (PD) or death from any cause.
Progression Free Survival (PFS) | Every 2 cycles,up to 24 months (each cycle is 28 days)
  The period of time between the start of the subject's first dose of medication and the first observation of disease progression (based on imaging) or the occurrence of death due to any cause.
Overall Survival (OS) | Cycle 1 Day 1 up to 24 months(each cycle is 28 days)
  Defined as the time between the date of first dose and death from any cause. Subjects who are alive as of the date of analysis will use and the date they last achieved survival as the cutoff time.
Plasma Concentration | Cycle 1 Day 1，Cycle 1 Day14，Cycle 1 Day 28 (each cycle is 28 days)
  PK samples of some subjects treated with study drugs will be collected for pharmacokinetic analysis in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Xingya Li, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (10):
- China (10):
  - The First Affiliated Hospital of Bengbu Medicaal University, Bengbu, Anhui
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Xuancheng People´s Hospital, Xuancheng, Anhui
  - Anyang Cancer Hospital, Anyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Nanjing Chest Hospital, Nanjing, Jiangsu
  - Sir Run Run Shaw Hospital (SRRSH),affiliated with Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Hospital Of Jiaxing, Jiaxing, Zhejiang